CLINICAL TRIAL: NCT01147068
Title: A Two-Part Placebo-Controlled Evaluation of the Safety and Immunogenicity of an A/Indonesia/5/05 Recombinant Hemagglutinin Influenza H5N1 Vaccine With and Without Glucopyranosyl Lipid A (GLA-SE) in Healthy Adults 18-49
Brief Title: Safety and Immunogenicity of PanBlok Influenza Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Responsible Party: Principal Investigator, Manon M.J. Cox, CEO, Protein Sciences Corporation
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSC22 GLA-SE
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Results first posted 2012-11-26 (Estimated); Last update posted 2012-11-26 (Estimated); Status verified 2012-10

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Injections, Intramuscular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- PanBlok 135µg No Adjuvant (Experimental): 135µg recombinant hemagglutinin, no adjuvant; Two 0.5 mL IM injections 21 days apart
  Interventions: Biological: 0.5mL Intramuscular Injection
- PanBlok 45µg No Adjuvant (Experimental): 45µg recombinant hemagglutinin, no adjuvant; Two 0.5 mL IM injections 21 days apart
  Interventions: Biological: 0.5mL Intramuscular Injection
- PanBlok 45µg and GLA 1.0µg, SE 2% (Experimental): 45µg recombinant hemagglutinin and Glucopyranosyl Lipid A 1.0µg in a 2% oil-in-water stable emulsion; Two 0.5 mL IM injections 21 days apart
  Interventions: Biological: 0.5mL Intramuscular Injection
- PanBlok 15µg and GLA 1.0µg, SE 2% (Experimental): 15µg recombinant hemagglutinin and Glucopyranosyl Lipid A 1.0µg in a 2% oil-in-water stable emulsion; Two 0.5 mL IM injections 21 days apart
  Interventions: Biological: 0.5mL Intramuscular Injection
- PanBlok 7.5µg and GLA 1.0µg, SE 2% (Experimental): 7.5µg recombinant hemagglutinin and Glucopyranosyl Lipid A 1.0µg in a 2% oil-in-water stable emulsion; Two 0.5 mL IM injections 21 days apart
  Interventions: Biological: 0.5mL Intramuscular Injection
- PanBlok 3.8µg and GLA 1.0µg, SE 2% (Experimental): 3.8µg recombinant hemagglutinin and Glucopyranosyl Lipid A 1.0µg in a 2% oil-in-water stable emulsion; Two 0.5 mL IM injections 21 days apart
  Interventions: Biological: 0.5mL Intramuscular Injection
- Placebo (Placebo Comparator): 0.9% Sodium Chloride; Two 0.5 mL IM injections 21 days apart
  Interventions: Biological: 0.5mL Intramuscular Injection

INTERVENTIONS:
Biological: 0.5mL Intramuscular Injection — 0.5mL intramuscular injection on day 0 and day 21 in the deltoid muscle
  Other Names: rHA; recombinant hemagglutinin; PanBlok

SUMMARY:
The purpose of this study is to investigate the safety and immunogenicity of a recombinant hemagglutinin (rHA) influenza vaccine derived from A/Indonesia/05/2005 (H5N1) administered at 4 dose levels in adjuvanted (GLA-SE) rHA formulations and 2 dose levels in unadjuvanted rHA formulations.

DETAILED DESCRIPTION:
All currently licensed influenza vaccines in the United States are produced in embryonated hen's eggs. There are several well-recognized disadvantages to the use of eggs as the substrate for influenza vaccine. Eggs require specialized manufacturing facilities and could be difficult to scale up rapidly in response to an emerging need such as a pandemic. It is usually necessary to adapt candidate vaccine viruses for high-yield growth in eggs, a process that can be time consuming, is not always successful, and can select receptor variants that may have suboptimal immunogenicity. In addition, agricultural diseases that affect chicken flocks, and that might be an important issue in a pandemic due to an avian influenza virus strain, could easily disrupt the supply of eggs for vaccine manufacturing. Therefore, development of alternative substrates for influenza vaccine production has been identified as a high-priority objective.

One potential alternative method for production of influenza vaccine is expression of the influenza virus hemagglutinin (HA) using recombinant DNA techniques. This alternative avoids dependence on eggs and is very efficient because of the high levels of protein expression under the control of the baculovirus polyhedrin promoter.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-49 years.
* Give written informed consent to participate.
* Healthy, as determined by medical history, physical examination, vital signs, and clinical safety laboratory evaluation
* Females should fulfill one of the following criteria:

  * At least one year post-menopausal;
  * Surgically sterile;
  * Will use oral, implantable, transdermal or injectable contraceptives for 30 days prior to first vaccination and until 28 days after the booster vaccination; or
  * Willing to use another reliable form of contraception approved by the Investigator (e.g., intrauterine device (IUD), female condom, diaphragm with spermicide, cervical cap, use of condom by the sexual partner or a sterile sexual partner) for 30 days prior to first vaccination and until 28 days after the booster vaccination.
* Women of childbearing potential must have a negative urine pregnancy test within 24 hours preceding receipt of first and booster vaccinations
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.

Exclusion Criteria:

* Persons under 18 years old or 50 years or older
* Persons with chronic illnesses such as cancer, diabetes, liver or kidney disease
* Persons taking medications or treatments that may adversely affect the immune system
* Persons with known allergy to eggs or other vaccine or adjuvant components
* Person currently pregnant, nursing mothers or planning a pregnancy within one month of vaccination
* Persons who have had a prior serious reaction to any influenza vaccine
* Persons with a known history of Guillain-Barré Syndrome
* Persons with a history of anaphylactic-type reaction to injected vaccines
* Persons with a history of drug or chemical abuse in the year preceding the study
* Persons who previously received an H5N1 influenza vaccine or who plan to receive an H5N1 influenza vaccine while participating in the study
* Persons who received a seasonal influenza vaccine six months prior to enrollment (may delay enrollment)
* Persons who received any other vaccine within one week prior to enrollment (may delay enrollment)
* Persons who have had a respiratory illness or illness with fever within three days of study enrollment (may delay enrollment)
* Persons currently participating in another research study involving any study medications (investigational drugs or vaccines).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 392 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Treanor, MD, Principal Investigator — University of Rochester
Locations (4):
- United States (4):
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Meridian Clinical Research, Omaha, Nebraska
  - University of Rochester, Rochester, New York
  - Benchmark Research, Fort Worth, Texas

REFERENCES:
- [Derived] Treanor JJ, Essink B, Hull S, Reed S, Izikson R, Patriarca P, Goldenthal KL, Kohberger R, Dunkle LM. Evaluation of safety and immunogenicity of recombinant influenza hemagglutinin (H5/Indonesia/05/2005) formulated with and without a stable oil-in-water emulsion containing glucopyranosyl-lipid A (SE+GLA) adjuvant. Vaccine. 2013 Nov 19;31(48):5760-5. doi: 10.1016/j.vaccine.2013.08.064. Epub 2013 Sep 27. PMID 24075920
- See also: Related Info — http://proteinsciences.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults 18-49 years of age were screened in participating outpatient clinics for eligibility within 30 days of randomization during the 2010 influenza season.
Pre-assignment Details: Subjects whose laboratory values were exclusionary were not randomized. Women of child-bearing potential were required to have a negative pregnancy test.
Groups:
- Placebo: 0.9% Sodium Chloride; Two 0.5 mL IM injections 21 days apart
  0.5mL Intramuscular Injection : 0.5mL intramuscular injection on day 0 and day 21 in the deltoid muscle
- PanBlok 135µg No Adjuvant: 135µg recombinant hemagglutinin, no adjuvant; Two 0.5 mL IM injections 21 days apart
  0.5mL Intramuscular Injection : 0.5mL intramuscular injection on day 0 and day 21 in the deltoid muscle
- PanBlok 45µg No Adjuvant: 45µg recombinant hemagglutinin, no adjuvant; Two 0.5 mL IM injections 21 days apart
  0.5mL Intramuscular Injection : 0.5mL intramuscular injection on day 0 and day 21 in the deltoid muscle
- PanBlok 45µg and GLA 1.0µg, SE 2%: 45µg recombinant hemagglutinin and Glucopyranosyl Lipid A 1.0µg in a 2% oil-in-water stable emulsion; Two 0.5 mL IM injections 21 days apart
  0.5mL Intramuscular Injection : 0.5mL intramuscular injection on day 0 and day 21 in the deltoid muscle
- PanBlok 15µg and GLA 1.0µg, SE 2%: 15µg recombinant hemagglutinin and Glucopyranosyl Lipid A 1.0µg in a 2% oil-in-water stable emulsion; Two 0.5 mL IM injections 21 days apart
  0.5mL Intramuscular Injection : 0.5mL intramuscular injection on day 0 and day 21 in the deltoid muscle
- PanBlok 7.5µg and GLA 1.0µg, SE 2%: 7.5µg recombinant hemagglutinin and Glucopyranosyl Lipid A 1.0µg in a 2% oil-in-water stable emulsion; Two 0.5 mL IM injections 21 days apart
  0.5mL Intramuscular Injection : 0.5mL intramuscular injection on day 0 and day 21 in the deltoid muscle
- PanBlok 3.8µg and GLA 1.0µg, SE 2%: 3.8µg recombinant hemagglutinin and Glucopyranosyl Lipid A 1.0µg in a 2% oil-in-water stable emulsion; Two 0.5 mL IM injections 21 days apart
  0.5mL Intramuscular Injection : 0.5mL intramuscular injection on day 0 and day 21 in the deltoid muscle
Period: Subjects That Received 1st Dose
Arm/Group | Placebo | PanBlok 135µg No Adjuvant | PanBlok 45µg No Adjuvant | PanBlok 45µg and GLA 1.0µg, SE 2% | PanBlok 15µg and GLA 1.0µg, SE 2% | PanBlok 7.5µg and GLA 1.0µg, SE 2% | PanBlok 3.8µg and GLA 1.0µg, SE 2%
Started | 60 | 57 | 55 | 56 | 56 | 53 | 55
Completed | 60 | 57 | 55 | 56 | 56 | 53 | 55
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Subjects That Received 2nd Dose
Arm/Group | Placebo | PanBlok 135µg No Adjuvant | PanBlok 45µg No Adjuvant | PanBlok 45µg and GLA 1.0µg, SE 2% | PanBlok 15µg and GLA 1.0µg, SE 2% | PanBlok 7.5µg and GLA 1.0µg, SE 2% | PanBlok 3.8µg and GLA 1.0µg, SE 2%
Started | 60 | 57 | 55 | 56 | 56 | 53 | 55
Completed | 59 | 52 | 52 | 56 | 55 | 51 | 55
Not Completed | 1 | 5 | 3 | 0 | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Ineligible | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Did not complete the study | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 3 | 3 | 0 | 1 | 0 | 0
Period: Subjects That Completed Safety Follow-up
Arm/Group | Placebo | PanBlok 135µg No Adjuvant | PanBlok 45µg No Adjuvant | PanBlok 45µg and GLA 1.0µg, SE 2% | PanBlok 15µg and GLA 1.0µg, SE 2% | PanBlok 7.5µg and GLA 1.0µg, SE 2% | PanBlok 3.8µg and GLA 1.0µg, SE 2%
Started | 60 (Participants were eligible for follow-up regardless of number of doses received.) | 57 (One subject was ineligible, one subject did not complete the study, and the other data is unknown.) | 55 (Data on three subjects is unknown.) | 56 | 56 (Data for one subject is unknown.) | 53 (One subject was lost to follow up and one subject did not complete the study.) | 55
Completed | 59 | 56 | 55 | 54 | 56 | 52 | 54
Not Completed | 1 | 1 | 0 | 2 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PanBlok 135µg No Adjuvant | PanBlok 45µg No Adjuvant | PanBlok 45µg and GLA 1.0µg, SE 2% | PanBlok 15µg and GLA 1.0µg, SE 2% | PanBlok 7.5µg and GLA 1.0µg, SE 2% | PanBlok 3.8µg and GLA 1.0µg, SE 2% | Total
Number analyzed (Participants) | 60 | 57 | 55 | 56 | 56 | 53 | 55 | 392
Age Continuous [Median (Full Range); unit: years] — The median was measured based on the total population of each arm.
  years | 32.0 [18 to 49] | 30.0 [18 to 48] | 32.0 [18 to 49] | 31.0 [18 to 49] | 33.5 [18 to 49] | 27.0 [19 to 48] | 33.0 [19 to 49] | 32.2 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 35 | 32 | 30 | 43 | 34 | 25 | 232
  Male | 27 | 22 | 23 | 26 | 13 | 19 | 30 | 160

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Immunogenicity Measured by Seroconversion Rates of PanBlok With and Without Adjuvant Compared to Placebo in Healthy Adults 18-49 Years of Age.
Description: Immunogenicity was assessed by measuring the percentage of subjects in each group exhibiting seroconversion on Day 42. The treatment groups that received adjuvanted rHA were evaluated against non-adjuvanted rHA and placebo groups for whether they demonstrated seroconversion rates and 95% confidence intervals that met regulatory criterion for licensure.
Time Frame: 42 Days
Population: All randomized subjects who received study vaccine and had Day 0 and Day 42 efficacy data. The analysis results are generated by Southern Research Institute on the intention to treat efficacy population using whole virus.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PanBlok 135µg No Adjuvant | PanBlok 45µg No Adjuvant | PanBlok 45µg and GLA 1.0µg, SE 2% | PanBlok 15µg and GLA 1.0µg, SE 2% | PanBlok 7.5µg and GLA 1.0µg, SE 2% | PanBlok 3.8µg and GLA 1.0µg, SE 2%
Number analyzed (Participants) | 57 | 54 | 54 | 54 | 56 | 53 | 53
percentage of participants | 0 [0 to 0] | 32 [21 to 45] | 15 [8 to 27] | 82 [69 to 90] | 75 [62 to 84] | 66 [53 to 77] | 72 [58 to 82]

2. Secondary Outcome: Evaluation and Comparison of Immunogenicity From Geometric Mean Titers of PanBlok With and Without Adjuvant and Placebo in Healthy Adults 18-64 Years of Age.
Description: Immunogenicity was assessed by measuring the proportion of subjects that exhibited a geometric mean titer change from Day 0 to Day 42. The geometric mean titers from the PanBlok groups (with and without adjuvant)and placebo group were then compared.
Time Frame: Day 0, and Day 42
Population: All randomized subjects who received study vaccine and had Day 0 and Day 42 geometric mean titers. Analysis of results were generated by Southern Research Institute on the overall population using whole virus.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | PanBlok 135µg No Adjuvant | PanBlok 45µg No Adjuvant | PanBlok 45µg and GLA 1.0µg, SE 2% | PanBlok 15µg and GLA 1.0µg, SE 2% | PanBlok 7.5µg and GLA 1.0µg, SE 2% | PanBlok 3.8µg and GLA 1.0µg, SE 2%
Number analyzed (Participants) | 57 | 54 | 54 | 54 | 56 | 53 | 53
titer
  Day 0 | NA [NA to NA] — Titer was below limit of detection | NA [NA to NA] — Titer was below limit of detection | NA [NA to NA] — Titer was below limit of detection | NA [NA to NA] — Titer was below limit of detection | NA [NA to NA] — Titer was below limit of detection | NA [NA to NA] — Titer was below limit of detection | NA [NA to NA] — Titer was below limit of detection
  Day 42 | NA [NA to NA] — Titer was below limit of detection | 16.7 [12 to 24] | 10.7 [8 to 14] | 128.4 [93 to 177] | 94.5 [63 to 142] | 68.7 [45 to 104] | 71.7 [47 to 108]

3. Secondary Outcome: Serologic Response Rates at Day 21 Using PanBlok With and Without Adjuvant and Placebo in Healthy Adults 18-64 Years of Age
Description: Immunogenicity was assessed by measuring the seroconversion rates of subjects from Day 0 to Day 21 to determine and evaluate the immune response following a single dose of study vaccine. The results were compared using PanBlok with and without adjuvant and placebo in healthy adults
Time Frame: 21 Days
Population: All randomized subjects with Day 0 and Day 21 data analyzed by Cincinnati Children's Hospital Medical Center using the intent to treat population and CBER antigen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | PanBlok 135µg No Adjuvant | PanBlok 45µg No Adjuvant | PanBlok 45µg and GLA 1.0µg, SE 2% | PanBlok 15µg and GLA 1.0µg, SE 2% | PanBlok 7.5µg and GLA 1.0µg, SE 2% | PanBlok 3.8µg and GLA 1.0µg, SE 2%
Number analyzed (Participants) | 60 | 56 | 54 | 56 | 56 | 52 | 55
percentage of participants | 3 [0.4 to 11.5] | 4 [0.4 to 12.3] | 4 [0.5 to 12.7] | 11 [4 to 21.9] | 7 [2 to 17.3] | 8 [2.1 to 18.5] | 2 [0 to 9.7]

ADVERSE EVENTS:
Time Frame: All Adverse Events - 28 days following immunization; Serious adverse events, adverse events of special interest, and new onset of chronic illnesses for duration of 12-month follow-up after immunization.
Arm/Group | Placebo | PanBlok 135µg No Adjuvant | PanBlok 45µg No Adjuvant | PanBlok 45µg and GLA 1.0µg, SE 2% | PanBlok 15µg and GLA 1.0µg, SE 2% | PanBlok 7.5µg and GLA 1.0µg, SE 2% | PanBlok 3.8µg and GLA 1.0µg, SE 2%
Serious Adverse Events (participants affected / at risk) | 1/60 | 2/57 | 1/55 | 1/56 | 2/56 | 0/53 | 3/55
Other Adverse Events (participants affected / at risk) | 39/60 | 36/57 | 33/55 | 35/56 | 40/56 | 32/53 | 38/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | PanBlok 135µg No Adjuvant (N=57) | PanBlok 45µg No Adjuvant (N=55) | PanBlok 45µg and GLA 1.0µg, SE 2% (N=56) | PanBlok 15µg and GLA 1.0µg, SE 2% (N=56) | PanBlok 7.5µg and GLA 1.0µg, SE 2% (N=53) | PanBlok 3.8µg and GLA 1.0µg, SE 2% (N=55)
Worsening of Right Ankle Instability (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional Hernia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominopelvic Mass (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured/Cracked Vertebrae (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Intrauterine Fetal Demise (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Costochondritis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Left Upper Lobe Lung Nodule with Organizing Abscess (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Ovarian Cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pinched nerve between C3-6 (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-operative Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unspecified Protein Calorie Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=60) | PanBlok 135µg No Adjuvant (N=57) | PanBlok 45µg No Adjuvant (N=55) | PanBlok 45µg and GLA 1.0µg, SE 2% (N=56) | PanBlok 15µg and GLA 1.0µg, SE 2% (N=56) | PanBlok 7.5µg and GLA 1.0µg, SE 2% (N=53) | PanBlok 3.8µg and GLA 1.0µg, SE 2% (N=55)
Blood Cholesterol Increased (Blood and lymphatic system disorders) | 6 (6) | 4 (4) | 7 (7) | 5 (5) | 5 (5) | 3 (3) | 9 (9)
Alanine Aminotransferase Increased (Hepatobiliary disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 5 (5) | 3 (3)
Aspartate Aminotransferase Increased (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 4 (4)
Blood Glucose Increased (Investigations) | 4 (4) | 5 (5) | 4 (4) | 4 (4) | 4 (4) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 4 (4) | 0 (0)
Mean Cell Haemoglobin Concentration Decreased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 5 (5) | 1 (1) | 1 (1)
Carbon Dioxide Decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Gamma-Glutamyltransferase Increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Haemoglobin Decreased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Neutrophil Count Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Oropharngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
White Blood Cell Count Increased (Investigations) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 3 (3)
Blood Creatinine Increased (Investigations) | 5 (5) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Blood Urea Nitrogen/Creatinine Ratio Decreased (Investigations) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Haematocrit Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood Cholesterol Increased (Investigations) | 6 (6) | 4 (4) | 7 (7) | 5 (5) | 5 (5) | 3 (3) | 9 (9)
Haematocrit Increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Joint Sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Red Cell Distribution Width Increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The absence of a treatment group receiving a SE- or GLA-alone adjuvanted vaccine formulation is a limitation to the study conclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No